CLINICAL TRIAL: NCT06776705
Title: A Pilot Randomized Controlled Trial of MRI-guided Focused Low-intensity Transcranial Ultrasound Stimulation (TUS) for Sleep Disturbances in Patients With Chronic Tinnitus
Brief Title: Low-intensity TUS for Sleep Disturbances in Patients With Chronic Tinnitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, LU Hanna, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023.636
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-01

CONDITIONS: Tinnitus; Sleep Disturbances; Cognition
Keywords: Tinnitus; Cognitive Dysfunction; Sleep distubances; Transcranial ultrasound stimulation; Hippocampus; Complex attention; Simulation; Central Nervous System Diseases
MeSH Terms: conditions — Tinnitus; Parasomnias; Cognitive Dysfunction; Central Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active TUS (Active Comparator): In active TUS group, participants will receive 500 kHz low-intensity TUS.
  Interventions: Device: Low-intensity transcranial ultrasound stimulation
- Sham TUS (Sham Comparator): In sham TUS group, participants will not receive low-intensity TUS.
  Interventions: Device: Low-intensity transcranial ultrasound stimulation

INTERVENTIONS:
Device: Low-intensity transcranial ultrasound stimulation — Low-intensity TUS, as an advanced modality of transcranial brain stimulation, enables to stimulate the deep brain structures with optimized focality and specific frequency.

SUMMARY:
Background: Tinnitus, as a common symptom, can jeopardize the sleep quality and brain function and even lead to hearing loss and cognitive decline in elderly patients. The co-occurring tinnitus and sleep disturbances can significantly affect the cognitive functions and quality of life, and even be implicated as a key contributing factor in the development of prodromal dementia. At present, very few non-pharmacological therapies are developed for managing these comorbidities in elderly patients. Focused low-intensity transcranial ultrasound stimulation (TUS) enables to stimulation the deep brain structures, such as hippocampus, with optimized focality and specific frequency.

Objectives: We aim to 1) investigate the safety, feasibility and efficacy of a 2-week focused low-intensity TUS on the severity of tinnitus and sleep disturbances in elderly patients; 2) determine the sample size of a full-scale randomized clinical trial of low-intensity TUS in patients with tinnitus; 3) evaluate the effects of low-intensity TUS on the severity of tinnitus, sleep quality and cognitive functions at 2, 4 and 6 weeks after the treatments.

Design: A 2-week randomized, double-blind, controlled clinical trial. Methods: Chinese right-handed tinnitus patients with sleep disturbances (aged from 60 to 90 years) will be randomly assigned to a 2-week intervention of either low intensity TUS or sham TUS, with 7 participants per arm. Before intervention, T1-weighted magnetic resonance imaging (MRI) and diffusion-weighted imaging (DWI) data is used to construct individual realistic head model. Comprehensive assessments, including sleep quality, cognitive performance and quality of life will be conducted at baseline, 2nd week, 4th week and 6th week. Program adherence and adverse effects will be monitored throughout intervention.

DETAILED DESCRIPTION:
Significance: This study aims to investigate the feasibility, safety and efficacy of low intensity TUS for sleep disturbances in patients with tinnitus. It wills also test the program adherence, tolerability and adverse effects of this innovative neurotechnology. Information will be helpful for in-depth understanding the relationship of "tinnitus, sleep and cognition" and guiding the further studies of otology, sleep medicine and age-related neurodegenerative diseases.

Data analysis: The primary outcomes will be the changes in tinnitus symptoms and sleep quality, and the comparisons of group differences across different time points. Secondary outcomes will be the changes of cognitive functions and quality of life. Intention-to-treat analysis will be carried out. Changes of efficacy indicators from baseline to each follow up point will be tested with mixed effect model.

ELIGIBILITY:
Inclusion Criteria:

* Chinese, right-handed, aged from 60 to 80 years.
* Chronic tinnitus is defined as tinnitus with a duration of at least 3 months. Depending on the justification, different time course definitions of chronic tinnitus are possible.
* Sleep disturbances are defined as a Pittsburgh Sleep Quality Index (PSQI) total score above 5.
* No interference with independence in everyday activities.

Exclusion Criteria:

* Diseases of ear canal and tympanic membrane checked by otoscopic examination.
* Previous diagnosis of Meniere's disease and acoustic neuromas.
* Past history of neurological or mental disorders.
* Physically frail affecting attendance to treatment sessions.
* Already attending regular treatments, such as cognitive behavioral therapy or music therapy.
* Taking a psychotropic or other medication known to affect hearing functions.
* Significant communicative impairments.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Tinnitus Primary Functions Questionnaire (TPFQ) | 12 weeks
  A short 12-item version of TPFQ is used in this study. In the 12-item version, questions 7, 11, and 15 were chosen for concentration; questions 4, 8, and 10 were chosen for emotion; questions 2, 14, and 17 were chosen for hearing; and questions 16, 18, and 20 were chosen for sleep.
Pittsburg Sleep Quality Index (PSQI) | 12 weeks
  The PSQI is a 19-item questionnaire that includes seven areas of subjective sleep quality and patterns in adults over the last month including the following components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, SDs, use of sleeping medications, and daytime dysfunction. Each item in the scale is scored from 0 to 3 scale (0 = no difficulty; 3 = severe difficulty). The scores are added to yield a global score ranging from 0 to 21 (0 = no difficulty; 21 = severe difficulties in all areas). This scale has good reliability and validity psychometrics and is widely used in research: Cronbach's alpha (0.77 to 0.83), sensitivity (89.6%), specificity (86.5%)(Buysse et al., 1988). Greater score of PSQI indicates worse sleep quality.

SECONDARY OUTCOMES:
Tinnitus Handicap Inventory (THI) | 12 weeks
  THI is used to identify, quantify and evaluate the difficulties that patients with chronic tinnitus may experience in daily life. There are 25 items covering three aspects: functional, emotional and catastrophic. The THI score ranges from 0 to 100, with higher scores indicating more severe tinnitus burden and a seven-point change representing a minimal clinically important difference.
Attention network test (ANT) | 12 weeks
  Complex attention is measured by ANT. Within ANT paradigm, there are four types of cues: no cue, center cue, double cue, and spatial cue; and three types of ﬂankers: neutral, congruent, and incongruent. In a given trial, a central cross-ﬁxation point presents 400 to 1,600 ms (randomized), subsequently is replaced for 100 ms by one of four warning cues. The target, a central arrow, could appear above or below the cross-ﬁxation and is surrounded by two ﬂankers on each side.
Word-list learning test (WLLT) | 12 weeks
  WLLT, consisting of ten semantically non-associated words that is presented consecutively over three free trials of immediate recall, a 20-min delayed recall (to prevent recency effects).

CONTACTS AND LOCATIONS:
Overall Officials: Hanna LU, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Tai Po Hospital, Hong Kong, Hong Kong
  - Tai Po Hospital, Hong Kong, Tai Po District

IPD SHARING:
Plan to Share IPD: No
The data collected in this study may include the healthy information and medical records.

REFERENCES:
- [Derived] Ni X, Yuen YS, Li Z, Wang K, Yang NS, Yuan Y, Meng L, Guo L, Lu H. Focused low-intensity hippocampal transcranial ultrasound stimulation (TUS) for sleep disturbances in patients with chronic tinnitus: A study protocol for a pilot randomized controlled trial. PLoS One. 2025 Aug 6;20(8):e0329950. doi: 10.1371/journal.pone.0329950. eCollection 2025. PMID 40768410